CLINICAL TRIAL: NCT03201822
Title: Intake-dependent Effect of Cocoa Flavanol Absorption, Metabolism and Excretion in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Mars, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 429275
Record Dates: First submitted 2017-06-19; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: flavanol; ADME; cocoa flavanols; polyphenols

STUDY DESIGN:
Intervention Model Description: Randomized, double-masked and cross-over dietary intervention study in healthy young adult males
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 100 mg of Cocoa Flavanols/70 kg BW (Experimental): Fruit flavored non-dairy drink containing 100 cocoa flavanol/70 kg BW
  Interventions: Other: 100 mg of Cocoa Flavanols/70 kg BW
- 200 mg of Cocoa Flavanols/70 kg BW (Experimental): Fruit flavored non-dairy drink containing 200 cocoa flavanol/70 kg BW
  Interventions: Other: 200 mg of Cocoa Flavanols/70 kg BW
- 400 mg of Cocoa Flavanols/70 kg BW (Experimental): Fruit flavored non-dairy drink containing 400 cocoa flavanol/70 kg BW
  Interventions: Other: 400 mg of Cocoa Flavanols/70 kg BW
- 1000 mg of Cocoa Flavanols/70 kg BW (Experimental): Fruit flavored non-dairy drink containing 1000 cocoa flavanol/70 kg BW
  Interventions: Other: 1000 mg of Cocoa Flavanols/70 kg BW

INTERVENTIONS:
Other: 100 mg of Cocoa Flavanols/70 kg BW — Fruit-flavored non-dairy drink containing 100 cocoa flavanols/70kg BW.
  Arms: 100 mg of Cocoa Flavanols/70 kg BW
Other: 200 mg of Cocoa Flavanols/70 kg BW — Fruit-flavored non-dairy drink containing 200 cocoa flavanols/70kg BW.
  Arms: 200 mg of Cocoa Flavanols/70 kg BW
Other: 400 mg of Cocoa Flavanols/70 kg BW — Fruit-flavored non-dairy drink containing 400 cocoa flavanols/70kg BW.
  Arms: 400 mg of Cocoa Flavanols/70 kg BW
Other: 1000 mg of Cocoa Flavanols/70 kg BW — Fruit-flavored non-dairy drink containing 1000 cocoa flavanols/70kg BW.
  Arms: 1000 mg of Cocoa Flavanols/70 kg BW

SUMMARY:
A randomized, double-masked and cross-over dietary intervention study in healthy young adult males to evaluate the concentration of F-derived metabolites in plasma and urine after single acute intakes of F-containing drinks on four different test days.

DETAILED DESCRIPTION:
Flavanols (F) are plant-derived compounds commonly present in the human diet. Examples of F-containing foods and beverages are apples, chocolate, tea, wine, berries, pomegranate and nuts. The consumption of F-containing foods and beverages has been associated with improvements in cardiovascular health. In this context, there exists a great interest in describing the absorption, metabolism and excretion of F in humans, as it is thought that F-derived metabolites present in circulation are the mediators of F-beneficial effects in humans. Recently, we described a series of F-derived metabolites in circulation that are present after the consumption of a single acute intake amount of F in humans. A key question, however, is if the metabolites we observed after a single acute feeding are the same as those that occur in individuals who consume F-rich diets on a regular basis. Studies investigating the metabolism of numerous other xenobiotics have shown that the profile of metabolites can greatly vary over time, as well as with the amount of xenobiotic ingested. In this context, and considering that i) the amount of F-consumed from diet greatly varies among individuals, ii) recent epidemiology studies indicate that the vascular protective effects of F diets primarily occur when daily intake of F are relatively high; and iii) there is evidence of an intake amount-dependency on the vascular effects of F in dietary intervention studies; we submit it is important to assess whether or not there are F intake amount-dependent effects on the levels and profile of F-derived metabolites in humans. This study will provide new information concerning the F-derived metabolites that may be responsible for mediating F-beneficial effects in humans. We suggest the information that will be obtained from the outlined work will be particularly timely given ongoing discussion concerning the possible generation of dietary recommendations for F-rich foods.

ELIGIBILITY:
Inclusion Criteria:

* No prescription medications
* BMI 18.5 - 29.9 kg/m2
* Weight ≥ 110 pounds
* previously consumed cocoa and peanut products, with no adverse reactions

Exclusion Criteria:

* Adults unable to consent
* Prisoners
* Non-English speaking*
* BMI ≥ 30 kg/m2
* Allergies to nuts, cocoa and chocolate products
* Active avoidance of coffee and caffeinated soft drinks
* Under current medical supervision
* A history of cardiovascular disease, stroke, renal, hepatic, or thyroid disease
* History of clinically significant depression, anxiety or other psychiatric condition
* History of Raynaud's disease
* History of difficult blood draws
* Indications of substance or alcohol abuse within the last 3 years
* Current use of herbal, plant or botanical supplements (multi-vitamin/mineral supplements are allowed)
* Blood Pressure > 140/90 mm Hg
* GI tract disorders, previous GI surgery (except appendectomy)
* Self-reported malabsorption (e.g. difficulty digesting or absorbing nutrients from food, potentially leading to bloating, cramping or gas)
* Diarrhea within the last month, or antibiotic intake within the last month
* Vegetarian, Vegan, food faddists, individuals using non-traditional diets, on a weight loss diet or individual following diets with significant deviations from the average diet
* Metabolic panel results or complete blood counts that are outside of the normal reference range and are considered clinically relevant by the study physician
* Screening LDL ≥ 190 mg/dl for those who have 0-1 major risk factors apart from LDL cholesterol (i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL)
* Screening LDL ≥ 160 mg/dl for those who have 2 major risk factors apart from LDL cholesterol (i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL).

(using NCEP calculator http://hp2010.nhlbihin.net/atpiii/calculator.asp?usertype=prof)

* Screening LDL ≥ 130 mg/dl for those who have 2 major risk factors apart from LDL cholesterol (i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL), and a Framingham 10-year Risk Score 10-20% (Framingham risk calculated using NCEP calculator http://hp2010.nhlbihin.net/atpiii/calculator.asp?usertype=prof)
* Cold, flu, or upper respiratory condition at screening
* Currently participating in a clinical or dietary intervention study

Ages: 25 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2013-05-25 (Actual); Study Completion 2013-05-25 (Actual)

PRIMARY OUTCOMES:
Change in levels of gut microbiome derived metabolites in urine | Urine collected 12h previous to intervention and up to 24 h after intervention
  Gut microbiome derived metabolites include conjugates of 5-(3',4'-dihydroxyphenyl)-g-valerolatone metabolites
Change in levels of gut microbiome derived metabolites in plasma | Plasma collected before (0h) and up to 6h post intervention
  Gut microbiome derived metabolites include conjugates of 5-(3',4'-dihydroxyphenyl)-g-valerolatone
Change in levels of structurally related epicatechin metabolites in urine | Urine collected 12h previous to intervention and up to 24 h after intervention
  Structurally related epicatechin metabolites include sulfated, glucuronidated and/or methylated metabolites of epicatechin
Change in levels of structurally related epicatechin metabolites in plasma | Plasma collected before (0h) and up to 6h post intervention
  Structurally related epicatechin metabolites include sulfated, glucuronidated and/or methylated metabolites of epicatechin

SECONDARY OUTCOMES:
Composite of pharmacokinetic (PK) parameters of metabolites Maximum Plasma Concentration (CMax) | Before intervention (0h) and up to 24 h after intervention
  PK parameters: Cmax: maximum observed concentration in plasma;
Composite of pharmacokinetic (PK) parameters of metabolites Time to Maximum Plasma Concentration | Before intervention (0h) and up to 24 h after intervention
  tmax: time to maximum concentration in plasma;
Composite of pharmacokinetic (PK) parameters of metabolites Area Under the Curve | Before intervention (0h) and up to 24 h after intervention
  AUC0-t: area under the plasma concentration-time curve from hour 0 to the last measurable concentration in plasma;
Composite of pharmacokinetic (PK) parameters of metabolites Area Under the Curve extrapolated to infinity | Before intervention (0h) and up to 24 h after intervention
  AUC0-∞: area under the plasma concentration-time curve extrapolated to infinity;
Composite of pharmacokinetic (PK) parameters of metabolites Elimination Rate Constant | Before intervention (0h) and up to 24 h after intervention
  λZ: apparent terminal elimination rate constant in plasma;
Composite of pharmacokinetic (PK) parameters of metabolites Elimination Half-Life | Before intervention (0h) and up to 24 h after intervention
  t1/2: apparent terminal elimination half-life in plasma;
Composite of pharmacokinetic (PK) parameters of metabolites Systemic Clearance | Before intervention (0h) and up to 24 h after intervention
  CL/F: systemic clearance;
Composite of pharmacokinetic (PK) parameters of metabolites Renal Clearance | Before intervention (0h) and up to 24 h after intervention
  CLR: renal clearance;sampling interval and the total interval examined;
Composite of pharmacokinetic (PK) parameters of metabolites cumulative Amount Excreted in Feces | Before intervention (0h) and up to 24 h after intervention
  Aef(0-t): Cumulative amount excreted in the feces over each sampling interval and the total interval examined.
Composite of pharmacokinetic (PK) parameters of metabolites Volume of Distribution | Before intervention (0h) and up to 24 h after intervention
  Vd/F: apparent volume of distribution;
Composite of pharmacokinetic (PK) parameters of metabolites cumulative Amount Excreted in Urine | Before intervention (0h) and up to 24 h after intervention
  Aeu(0-t): cumulative amount excreted in the urine over each

CONTACTS AND LOCATIONS:
Overall Officials: Carl L Keen, PhD, Principal Investigator — UC Davis; Javier I Ottaviani, PhD, Study Director — Mars, Inc.
Locations (1):
- UC Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Only researchers listed in the protocol and approved by the IRB will have access to IPD.

REFERENCES:
- [Background] Schroeter H, Heiss C, Spencer JP, Keen CL, Lupton JR, Schmitz HH. Recommending flavanols and procyanidins for cardiovascular health: current knowledge and future needs. Mol Aspects Med. 2010 Dec;31(6):546-57. doi: 10.1016/j.mam.2010.09.008. Epub 2010 Sep 18. PMID 20854838
- [Background] Ottaviani JI, Momma TY, Kuhnle GK, Keen CL, Schroeter H. Structurally related (-)-epicatechin metabolites in humans: assessment using de novo chemically synthesized authentic standards. Free Radic Biol Med. 2012 Apr 15;52(8):1403-12. doi: 10.1016/j.freeradbiomed.2011.12.010. Epub 2011 Dec 23. PMID 22240152
- [Background] Koster H, Halsema I, Scholtens E, Knippers M, Mulder GJ. Dose-dependent shifts in the sulfation and glucuronidation of phenolic compounds in the rat in vivo and in isolated hepatocytes. The role of saturation of phenolsulfotransferase. Biochem Pharmacol. 1981 Sep 15;30(18):2569-75. doi: 10.1016/0006-2952(81)90584-0. No abstract available. PMID 6946775
- [Background] McCullough ML, Chevaux K, Jackson L, Preston M, Martinez G, Schmitz HH, Coletti C, Campos H, Hollenberg NK. Hypertension, the Kuna, and the epidemiology of flavanols. J Cardiovasc Pharmacol. 2006;47 Suppl 2:S103-9; discussion 119-21. doi: 10.1097/00005344-200606001-00003. PMID 16794446
- [Background] Heiss C, Kleinbongard P, Dejam A, Perre S, Schroeter H, Sies H, Kelm M. Acute consumption of flavanol-rich cocoa and the reversal of endothelial dysfunction in smokers. J Am Coll Cardiol. 2005 Oct 4;46(7):1276-83. doi: 10.1016/j.jacc.2005.06.055. PMID 16198843